CLINICAL TRIAL: NCT02235506
Title: A Comparison of Epidural Analgesia With Adding Sciatic Nerve Block to Continuous Femoral Nerve Block for Post-operative Pain Management Following Total Knee Arthroplasty
Brief Title: A Comparison of Epidural Block With Adding Sciatic Block to Continuous Femoral Block in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: apsj0901
Record Dates: First submitted 2014-09-01; First posted 2014-09-10 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epidural infusion (Experimental): In epidural infusion group, a lumbar epidural catheter was placed at the L3-4 level using loss-ofresistance procedure. ropivacaine 0.2% and fentayl 2mcg/ml were infused at a rate of 5ml/hr from the end of operation,
  Interventions: Procedure: epidural infusion; Device: epidural infusion
- femoral sciatic (Experimental): In femoral sciatic group, the femoral and sciatic nerve are located using ultrasound and 0.2% ropivacain is injected. A catheter is inserted to femoral nerve. From the end of operation, 0.2% ropivacaine was infused through the femoral catheter at a rate of 5ml/hr.
  Interventions: Procedure: femoral sciatic; Device: femoral sciatic

INTERVENTIONS:
Procedure: epidural infusion — Lumbar epidural catheter is placed at the L3-4 level using loss-ofresistance procedure. Fentayl 2mcg/ml and 0.2% ropivacaine are infused at a rate of 5ml/hr.
  Other Names: continuous lumbar epidural block
  Arms: epidural infusion
Procedure: femoral sciatic — After femoral and sciatic nerve are identified using ultrasound, 0.2% ropivacaine 20 mL is injected. A catheter is inserted to femoral nerve and 0.2% ropivacaine is infused through the femoral catheter at a rate of 5ml/hr from the end of surgery.
  Other Names: femoral nerve block and sciatic nerve block
  Arms: femoral sciatic
Device: epidural infusion — Lumbar epidural catheter is placed at the L3-4 level using loss-ofresistance procedure. Fentayl 2mcg/ml and 0.2% ropivacaine are infused at a rate of 5ml/hr.
  Other Names: perifix epidural catheter, B-Braoun
  Arms: epidural infusion
Device: femoral sciatic — After femoral and sciatic nerve are identified using ultrasound, 0.2% ropivacaine 20 mL is injected. A catheter is inserted to femoral nerve and 0.2% ropivacaine is infused through the femoral catheter at a rate of 5ml/hr from the end of surgery.
  Other Names: contiplex catheter and stimuplex needle; B-Braun
  Arms: femoral sciatic

SUMMARY:
The investigators compared continuous epidural infusion with combined continuous femoral and single-shot sciatic nerve blocks. The primary outcome was the incidence of side effects, and secondary outcomes were pain relief, motor blockade,morphine consumption, and rehabilitation indices.

DETAILED DESCRIPTION:
The parcicipants were randomly assingned to epidural infusion group and femoral sciatic block. In epidural infusion group, a lumbar epidural catheter was placed at the L3-4 level using loss-ofresistance procedure. ropivacaine 0.2% and fentayl 2mcg/ml were infused at a rate of 5ml/hr from the end of operation. In femoral sciatic group, the femoral and sciatic nerve are located using ultrasound and 0.2% ropivacain is injected. A catheter is inserted to femoral nerve. From the end of operation, 0.2% ropivacaine was infused through the femoral catheter at a rate of 5ml/hr. The incidence of side effects is measured.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification I-II
* total knee arthroplasty
* 18-90 years

Exclusion Criteria:

* allergic to the local anesthetics
* cognitive impairment such as dementia
* coagulopathy
* motor and sensory impairment
* patient refusal
* BMI >39

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of side effects | during 5 days after the end of operation
  Side effects: The patients were asked to their experience of dizziness, sedation, nausea/vomiting (PONV), and pruritus. Urinary retention: bladder volume was measured by ultrasonography and if the volume was more than 400 mL and if the patient was unable to void spontaneously, single catheterization was performed.

SECONDARY OUTCOMES:
Pain | during 5 days after the end of operation
  Pain according to visual analogue scale at rest and on mobilization.
Motor blockade at rest and on mobilization | during 5 days after the end of operation
  Motor blockade is estimated using a modified Bromage scale

CONTACTS AND LOCATIONS:
Overall Officials: Sangjin Park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Daegu, South Korea